CLINICAL TRIAL: NCT03008889
Title: A Feasibility Study of N-acetylcysteine for Self-injurious Behavior in Children With Autism Spectrum Disorder
Acronym: NAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Lawrence Scahill, MSN, PhD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00088115
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2020-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Repetitive Self-Injurious Behavior; N-acetylcysteine (NAC)
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants taking NAC (Experimental): Participants randomized to the active treatment study arm will receive gradually increasing doses of N-acetylcysteine (NAC) given as a dissolving tablet in juice or water. NAC is an over-the-counter oral dietary supplement that will be used a higher than usual doses in this study.
  Interventions: Drug: N-acetylcysteine
- Participants taking Placebo (Placebo Comparator): Participants randomized to placebo will receive dissolving tablets identical in size and appearance to the active treatment. Placebo capsules contain inactive ingredients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — Participants will start with taking 900mg of NAC once per day for one week (study days 1-7). At Day 7, parents (or primary caregiver) and subjects will return to the study site to review adverse events.
  In the absence of dose limiting adverse events attributable to the study drug, the dose will be gradually increased to 900 mg twice per day for study days 8-28.
  If this dose is well-tolerated, the dose will be increased to 900 three times per day for study days 29-63.
  Other Names: NAC
  Arms: Participants taking NAC
Drug: Placebo — Participants will start with taking 900mg of the placebo once per day for one week (study days 1-7). At Day 7, parents (or primary caregiver) and subjects will return to the study site to review adverse events. The dosing for the placebo will increase in the same fashion as the active treatment.
  In the absence of dose limiting adverse events attributable to the study drug, the dose will be gradually increased to 900 mg twice per day for study days 8-28.
  If this dose is well-tolerated, the dose will be increased to 900 three times per day for study days 29-63.
  Arms: Participants taking Placebo

SUMMARY:
The purpose of this study is to demonstrate the feasibility of a 9-week, randomized trial of N-acetylcysteine (NAC) compared to placebo in 14 children (age 5 to 12 years) with Autism Spectrum Disorder (ASD) and a moderate level of repetitive self-injurious behavior (SIB). Additional aims are to evaluate the positive predictive value of a screening method to classify children with automatically maintained self-injurious behavior; to evaluate the preliminary efficacy of NAC for reducing repetitive SIB in children with ASD; and to evaluate biomarkers and possible mechanisms of action of NAC in children with ASD.

DETAILED DESCRIPTION:
Self-injurious behavior (SIB) in children with autism spectrum disorder (ASD) can cause physical harm to the child and interfere with the child's ability to make use of educational programs and helpful treatments such as speech therapy. The turmoil caused by self-injurious behaviors in children with ASD invariably interferes with daily routines because family life often stops during these episodes and family members worry about setting off SIB between episodes. This project will use the detailed assessment methods developed in the field of behavior therapy to evaluate the potential for N-acetylcysteine (NAC) to treat children with ASD and moderate repetitive SIB. NAC is an over-the-counter dietary supplement that may have beneficial effects on the brain through its well-documented antioxidant effects and/or reduced glutamate signaling. In the proposed study, 14 children with ASD and repetitive SIB between the ages of 5 and 12 will be randomly assigned to gradually increasing doses of NAC or placebo for 9 weeks. The research team, parents and children will be blind to the treatment with NAC or placebo. Participants will come to the research site periodically to complete measures and behavioral assessments.

After the 9 weeks of treatment, children randomized to NAC who showed improvement will be encouraged to continue taking the supplement outside the study. Children who were randomly assigned to the placebo and showed no improvement will be offered open-label treatment with NAC. Children who did not improve while taking NAC or those who improved while on the placebo will be advised on next steps by the study team.

The goal of this feasibility study is establish the acceptability viability of study procedures in this vulnerable population, to learn about the potential benefits and adverse effects of NAC. Demonstrating these feasibility aims and the preliminary efficacy and safety of NAC is a prerequisite for planning a larger, more definitive, study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Autism Spectrum Disorder (ASD)
* Confirmed presence of moderate Self Injurious Behavior (SIB)
* Score > 16 on the parent-rated Aberrant Behavior Checklist Irritability subscale (moderate level of disruptive behavior)
* Classified as having automatically maintained SIB (determined during screening by a detailed functional analysis)

Exclusion Criteria:

* On a stable medication dose for less than 4 weeks
* Planned change in medication during the 9-week trial
* Had one or more seizures in the last 6 months

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Scahill, MSN, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were eight consented (or enrolled) participants. Out of the eight participants, one screened failed early, and seven subjects were eligible for the Screening method for classifying self-injurious behavior (SIB) before randomization. Out of those seven, 3 passed screening, and one of the 3 withdrew due to study burden. Two participants were randomized to an intervention (NAC or placebo).
Groups:
- Participants Taking NAC: Participants randomized to the active treatment study arm will receive gradually increasing doses of N-acetylcysteine (NAC) given as a dissolving tablet in juice or water. NAC is an over-the-counter oral dietary supplement that will be used a higher than usual doses in this study.
  N-acetylcysteine: Participants will start with taking 900mg of NAC once per day for one week (study days 1-7). At Day 7, parents (or primary caregiver) and subjects will return to the study site to review adverse events.
  In the absence of dose limiting adverse events attributable to the study drug, the dose will be gradually increased to 900 mg twice per day for study days 8-28.
  If this dose is well-tolerated, the dose will be increased to 900 three times per day for study days 29-63.
- Participants Taking Placebo: Participants randomized to placebo will receive dissolving tablets identical in size and appearance to the active treatment. Placebo capsules contain inactive ingredients.
  Placebo: Participants will start with taking 900mg of the placebo once per day for one week (study days 1-7). At Day 7, parents (or primary caregiver) and subjects will return to the study site to review adverse events. The dosing for the placebo will increase in the same fashion as the active treatment.
  In the absence of dose limiting adverse events attributable to the study drug, the dose will be gradually increased to 900 mg twice per day for study days 8-28.
  If this dose is well-tolerated, the dose will be increased to 900 three times per day for study days 29-63.
Period: Overall Study
Arm/Group | Participants Taking NAC | Participants Taking Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Taking NAC | Participants Taking Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 8 (0) | 9 (0) | 8.5 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Randomized
Description: Goal: randomize 1.75 participants per month
Time Frame: 12 months (throughout the duration of the study)
Measure: Number; unit: percentage of participants randomized
Groups:
- Participants Taking NAC: Participants randomized to the active treatment study arm received gradually increasing doses of N-acetylcysteine (NAC) given as a dissolving tablet in juice or water. NAC is an over-the-counter oral dietary supplement that was used at a higher than usual doses in this study.
  N-acetylcysteine: Participants started taking 900mg of NAC once per day for one week (study days 1-7). At Day 7, parents (or primary caregiver) and subjects returned to the study site to review adverse events.
  In the absence of dose limiting adverse events attributable to the study drug, the dose was gradually increased to 900 mg twice per day for study days 8-28.
  If this dose was well-tolerated, the dose was increased to 900 three times per day for study days 29-63.
- Participants Taking Placebo: Participants randomized to placebo received dissolving tablets identical in size and appearance to the active treatment. Placebo capsules contained inactive ingredients.
  Placebo: Participants started taking 900mg of the placebo once per day for one week (study days 1-7). At Day 7, parents (or primary caregiver) and subjects returned to the study site to review adverse events. The dosing for the placebo was increased in the same fashion as the active treatment.
  In the absence of dose limiting adverse events attributable to the study drug, the dose was gradually increased to 900 mg twice per day for study days 8-28.
  If this dose was well-tolerated, the dose was increased to 900 three times per day for study days 29-63.
Arm/Group | Participants Taking NAC | Participants Taking Placebo
Number analyzed (Participants) | 1 | 1
percentage of participants randomized | 100 | 100

2. Primary Outcome: Attrition Rate
Description: Attrition rate is defined as the percent of subjects who did not complete the study. Goal:less than 15% (to indicate that study was acceptable to participants and parents).
Time Frame: 12 months (throughout the duration of the study)
Measure: Number; unit: percentage of participants
Arm/Group | Participants Taking NAC | Participants Taking Placebo
Number analyzed (Participants) | 1 | 1
percentage of participants | 0 | 0

3. Primary Outcome: Study Medication Compliance
Description: Goal: at least 70% treatment compliance (tablet counts and drug dairies).
Time Frame: 12 months (throughout the duration of the study)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Taking NAC | Participants Taking Placebo
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

4. Primary Outcome: Successful Collection of Outcome Measures
Description: Goal: at least 80% collection of essential outcome data to demonstrate the feasibility of data collection procedures.
Time Frame: 12 months (throughout the duration of the study)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Taking NAC | Participants Taking Placebo
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

5. Primary Outcome: Parent Satisfaction Rating
Description: Goal: at least 80% of parents will agree or strongly agree when asked in an anonymous survey that they would recommend the study and the study treatment to other parents of children with ASD and SIB.
Time Frame: Week 9 (at the end of the study intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Taking NAC | Participants Taking Placebo
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

6. Secondary Outcome: Positive Predictive Value of Screening Method of Classifying Self-injurious Behavior (SIB) by Type.
Description: Goal: at least 75% positive predictive value of our screening method to classify children with automatically maintained self-injurious behavior using a semi-structured interview at screening compared to the findings of five- to six-hour functional analysis at baseline. Only children who appear to have automatically maintained SIB will be referred for the baseline evaluation.
  Demonstrating a high positive predictive value for the screening method is a necessary prerequisite for launching a larger study. Using the formula: Positive Predictive Value (PPV) = screen positive and true cases ÷ all positive screens, a value of 75% or greater would indicate success of the screening method used.
Time Frame: 12 months (duration of the study)
Population: Screening method for classifying self-injurious behavior (SIB) happened before randomization. Of the 8 participants that consented, one was excluded due to asthma. Results show participants that were classified with repetitive SIB.
Measure: Count of Participants; unit: Participants
Groups:
- Consented Participants Before Randomization: Participants consented in the trial, before randomization.
Arm/Group | Consented Participants Before Randomization
Number analyzed (Participants) | 7
Participants | 3

7. Secondary Outcome: Aberrant Behavior Checklist Irritability Subscale Score at Baseline and 9 Weeks Post-intervention
Description: The Aberrant Behavior Checklist (ABC) is a commonly used 58-item parent-rated measure of overall behavioral problems. The Irritability subscale is comprised of 15 items reflecting tantrums, aggression and self injury. Range is 0 to 45, higher scores indicate higher severity. As a preliminary efficacy outcome, it was calculated the average score at baseline and Week 9 post-intervention.
Time Frame: Baseline, Week 9
Measure: Number; unit: score on a scale
Arm/Group | Participants Taking NAC | Participants Taking Placebo
Number analyzed (Participants) | 1 | 1
score on a scale
  Score at Baseline | 31 | 28
  Score at 9-Weeks | 23 | 29

8. Secondary Outcome: Number of Self-Injurious Behavior Events
Description: Direct observation of the frequency of SIB was collected at baseline in a separate observational session after completing the functional analysis and again at Week 9. Investigators set a benchmark of an average decline in the frequency of SIB of 50% within the NAC group.
Time Frame: Baseline, Week 9
Measure: Number; unit: Self injurious events
Arm/Group | Participants Taking NAC | Participants Taking Placebo
Number analyzed (Participants) | 1 | 1
Self injurious events
  Baseline | 219 | 93
  9-Weeks | 59 | 655

9. Secondary Outcome: Change in Clinical Global Impression (CGI-I) Scale at 9 Weeks Post-intervention
Description: The Clinical Global Impression (CGI-I) scale is a 7-item scale from 1 (Very Much Improved) through 4 (No Change) to 7 (Very Much Worse). By convention, scores of 2 (Much Improved) or 1 (Very Much Improved) are used to define positive response.
Time Frame: Week 9
Measure: Number; unit: score on a scale
Arm/Group | Participants Taking NAC | Participants Taking Placebo
Number analyzed (Participants) | 1 | 1
score on a scale | 2 | 4

10. Secondary Outcome: Change in Biomarkers and Possible Mechanisms of Action of NAC in Children With ASD.
Description: Changes amino acid levels before and after NAC treatment: cysteine/cystine and glutathione/glutathione disulfide (GSH/GSSG) ratios (antioxidant effects), glutamate and glutamate/glutamine ratio (glutamate signaling) and GABA levels.
Time Frame: Baseline, Week 9
Population: Blood samples were collected and processed in accordance with the protocol. In consultation with our biochemist collaborator, we did not proceed with the multiple laboratory procedures to analyze the sample. Our collaborator indicated that the findings would not be interpretable because we only had two subjects.
Arm/Group | Participants Taking NAC | Participants Taking Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: Each subject was followed by two blinded clinicians. A treating clinician who monitored adverse events and managed the dose of the study medication. An independent evaluator assessed therapeutic response and did not discuss adverse events or medication dose with parent and child.
Arm/Group | Participants Taking NAC | Participants Taking Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Taking NAC (N=1) | Participants Taking Placebo (N=1)
Early morning awakening (General disorders) | 1 (1) | 0 (0)
Drowsiness (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased Appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight gain (General disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT03008889/Prot_SAP_000.pdf